CLINICAL TRIAL: NCT03621085
Title: Analgesics in the Pre-hospital Setting: Implications on Hemorrhage Tolerance - Ketamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: STU 092017-068
Record Dates: First submitted 2018-08-01; First posted 2018-08-08 (Actual); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Hemorrhage; Healthy
MeSH Terms: conditions — Hemorrhage | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Subjects will receive up to 20 mg Ketamine Hydrochloride while the effects of this drug on tolerance to a hemorrhagic insult will be assessed.
  Interventions: Drug: Ketamine Hydrochloride
- Placebo (Placebo Comparator): Subjects will receive placebo while the effects of this drug on tolerance to a hemorrhagic insult will be assessed.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine Hydrochloride — A total of 20 mg of Ketamine Hydrochloride will be administered intravenously
  Arms: Ketamine
Other: Placebo — Subjects will receive placebo
  Arms: Placebo

SUMMARY:
The purpose of this project is to test how ketamine, an analgesics currently employed in the pre-hospital setting by the US Army, alters the capacity to tolerate a hemorrhagic insult in humans.

DETAILED DESCRIPTION:
Pain management on the battlefield is critical for the wellbeing of the soldier. Given that a hemorrhagic injury on the battlefield is virtually always associated with pain, it is paramount that the selected pain medication does not disrupt appropriate physiological mechanisms that are beneficial towards the maintenance of blood pressure and vital organ blood flow during that hemorrhagic insult. Current guidelines for the selection of pain medications of a hemorrhaging soldier are based upon limited scientific evidence, with the vast majority of supporting studies being conducted on anesthetized animals. Thus, the interaction between hemorrhagic shock and pain medications commonly employed on the battlefield is yet to be determined in the conscious humans.

With this background, we will test the hypothesis that ketamine will impair the capacity for a conscious human to tolerate a hemorrhagic insult.

The obtained data will provide the necessary scientific evidence in humans to support the Committee on Tactical Combat Casualty Care (CoTCCC) guidelines on the analgesic of choice for moderate to severe injuries where the casualty is in hemorrhagic shock. Notably, such data will identify the analgesic that least compromises a human's ability to tolerate a hemorrhagic insult, ultimately providing critical information to the combat medic on which analgesic should be employed for such an injury.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* Healthy
* Non-obese (body mass index less than 30 kg/m2)
* Body mass greater than or equal to 65 kg

Exclusion Criteria:

* Subjects not in the defined age range
* Subjects who have cardiac, respiratory, neurological and/or metabolic illnesses
* Any known history of renal or hepatic insufficiency/disease
* Pregnancy or breast feeding
* Body mass less than 65 kg
* Current smokers, as well as individuals who regularly smoked within the past 3 years
* Positive urine drug screen
* Currently taking pain modifying medication(s)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: craig G Crandall, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watso JC, Huang M, Moralez G, Cramer MN, Hendrix JM, Cimino FA 3rd, Belval LN, Hinojosa-Laborde C, Crandall CG. Low dose ketamine reduces pain perception and blood pressure, but not muscle sympathetic nerve activity, responses during a cold pressor test. J Physiol. 2021 Jan;599(1):67-81. doi: 10.1113/JP280706. Epub 2020 Oct 20. PMID 33017047
- [Result] Huang M, Watso JC, Moralez G, Cramer MN, Hendrix JM, Yoo JK, Badrov MB, Fu Q, Hinojosa-Laborde C, Crandall CG. Low-dose ketamine affects blood pressure, but not muscle sympathetic nerve activity, during progressive central hypovolemia without altering tolerance. J Physiol. 2020 Dec;598(24):5661-5672. doi: 10.1113/JP280491. Epub 2020 Oct 20. PMID 33084081

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine First, Then Placebo: Ketamine visit (20 mg) first, then Placebo visit (saline)
- Placebo First, Then Ketamine: Placebo visit (saline) first, then Ketamine visit (20 mg)
Period: Enrollment
Arm/Group | Ketamine First, Then Placebo | Placebo First, Then Ketamine
Started | 22 | 21
Completed | 16 | 14
Not Completed | 6 | 7
Period: First Visit
Arm/Group | Ketamine First, Then Placebo | Placebo First, Then Ketamine
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0
Period: Washout (at Least 48 Hours)
Arm/Group | Ketamine First, Then Placebo | Placebo First, Then Ketamine
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0
Period: Second Visit
Arm/Group | Ketamine First, Then Placebo | Placebo First, Then Ketamine
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 33
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Stress Index
Description: Tolerance to a simulated hemorrhagic challenge will be assessed, for both the placebo and ketamine limbs, by causing progressive central hypovolemia via lower-body negative pressure (LBNP). This progressive lower-body negative pressure challenge will be performed until the onset of syncopal symptoms (defined as: profound bradycardia, a precipitous drop in arterial blood pressure and accompanying narrowing of pulse pressure, a sustained systolic blood pressure less than 80 mmHg, and/or subjective symptoms such as light-headedness, sweating, nausea, or dizziness). The primary variable will be the quantification of lower-body negative pressure that is required to cause these symptoms. This quantification will be objectively measured via a cumulative stress index which is calculated as the sum of the product of the LBNP level and the duration of each level, until test termination (i.e., 40 mmHg x 3 min + 50 mmHg x 3 min, etc).
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: mmHg x minutes
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 30 | 30
mmHg x minutes | 635 (391) | 649 (362)

2. Secondary Outcome: Pressure Pain Tolerance
Description: Pain assessments will be conducted using a digital algometer to obtain maximum pain thresholds caused by pressure. This pain assessment technique is conducted by applying the tip of a hand-held digital algometer on the subject's digit. Force is gradually increased and the peak force is recorded when the subject first reports a painful sensation. Removal of the pressure from the algometer immediately relieves the painful sensation and the subject can voluntarily stop the test at any time. This assessment will be performed after the subject has received placebo and ketamine.
Time Frame: 12 months
Population: Pressure pain tolerance was evaluated in a subset of individuals
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 20 | 20
Kilograms | 3.3 (1.0) | 1.6 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from until discharge from the final data collection visit, which typically occurred 6 to 12 months after consent/screening.
Description: Each participant completed both drug and placebo conditions, therefore, groups are combined for adverse event reporting.
Groups:
- Ketamine: Ketamine trials
- Placebo: Placebo trials
Arm/Group | Ketamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03621085/Prot_003.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT03621085/SAP_004.pdf
  • Informed Consent Form (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03621085/ICF_005.pdf